CLINICAL TRIAL: NCT02123797
Title: Building a Multidisciplinary Bridge Across the Quality Chasm in Thoracic Oncology
Status: Completed | Type: Observational
Sponsor: Baptist Memorial Health Care Corporation (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Raymond Osarogiagbon, MD, Director, Thoracic Oncology Research Group, Mutidisciplinary Program, Baptist Memorial Health Care Corporation
Other Study IDs: The Milestone Project
Record Dates: First submitted 2014-04-22; First posted 2014-04-28 (Estimated); Results first posted 2020-07-02 (Actual); Last update posted 2020-07-02 (Actual); Status verified 2020-06

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Multidisciplinary Clinic Patients: : 150 multidisciplinary clinic patients matched 1:2 with 300 serial care patients
- Serial Care Patients: 150 multidisciplinary clinic patients matched 1:2 with 300 serial care patients = 450 patients Since Baptist Health Care System manages >800 new cases each year, 300 of which are expected to be seen in multidisciplinary clinic, in practice, we conservatively expect to be able to recruit 150 cases from multidisciplinary clinic and 300 matched serial care controls (1:2 match) in 18 months.
- Multidisciplinary Caregivers: Consenting caregivers of consented multidisciplinary clinic patients (patients seen by multiple specialists at a single appointment time).
- Serial Care Caregivers: Consenting caregivers of consented serial care patients (patients who receive the current system of linear, sequential, referral-based care delivery).
- Clinical Providers: Clinical providers who referred at least 5 patients to the multidisciplinary program and consented to the study.

SUMMARY:
Lung cancer kills 160,000 patients annually; this represents 28% of all US cancer deaths. The overall year survival rate has only improved from 12% to 17% in 33 years. This failure reflects the innate lethality of lung cancer, but also reflects defects in patient care delivery. Care for the lung cancer patient starts with an abnormal radiologic scan, proceeds through a diagnostic biopsy, tests to determine the extent of spread of the disease (stage), selection of appropriate treatment, and finally ends with patient outcomes. At each step are multiple options and independent specialists, each one engaged by a process of sequential referrals in the serial care model. This process is often not user-friendly, is riddled with inefficiency, delays, and outcome variances.

The coordinated multidisciplinary model, in which patients and their doctors collaborate to provide evidence-based care, is believed by experts to be superior, but has few examples of successful implementation. The implementation gap exists because of the paucity of good quality data, and lack of implementation know-how.

Embedded in the highest US lung cancer mortality zone, the greater Memphis area has a racially, culturally, economically and geographically diverse population. The investigators research group has shown how poor quality care impairs patient survival in this region and in the greater US. The investigators have linked patient survival to compliance with multidisciplinary care plans. In this project, the investigators propose to rigorously test the impact of the multidisciplinary care model on patient outcomes in a community-based, private practice environment, similar to where 70% of lung cancer care is delivered in the US.

The objective of this study is to provide high-level evidence of the impact of multidisciplinary care on lung cancer patient outcomes. Multidisciplinary care is defined as a model of care in which patients, their care-givers and key specialists concurrently and directly evaluate the same patients in the presence of the patients and their informal caregivers, in order to develop evidence-based consensus care plans

DETAILED DESCRIPTION:
Within the Baptist Memorial Health Care system, the Multidisciplinary Thoracic Oncology Program has two components: Primarily, the program is centered in a multidisciplinary clinic, wherein patients and their informal caregivers are seen by multiple specialists at a single appointment time; secondarily, the program includes a multidisciplinary conference, wherein all of the specialists potentially involved in lung cancer care discuss patients referred for presentation and make consensus recommendations for care. This study focuses primarily on the experience and outcomes of care delivered to patients evaluated in the multidisciplinary clinic. However, data from the conference will also be included in some aspects of the study. The goal is to improve the access and quality of thoracic oncologic care delivery within the Baptist Healthcare System The investigators specific aim is to perform a prospective, matched cohort comparative effectiveness study of patients receiving serial vs. multidisciplinary care, with key patient-centered endpoints (survival, stakeholder satisfaction with the care experience, timeliness and stage-appropriateness of care, quality of staging). Serial care is defined as the current system of linear, sequential, referral-based care delivery.

ELIGIBILITY:
Inclusion Criteria:

- All patients who undergo care for lung cancer or an undiagnosed lung mass within the Baptist Memorial Health Care Corporation's hospitals from January 1, 2009 until the end of the defined study period will be eligible for inclusion in the data collection for this study. In addition, caregivers of patients within the same institution and within the study window, clinical care providers (doctors and nurses) who have taken care of patients within the eligible institutions during the study window.

Exclusion Criteria:

* Patients who do not have a radiology-identified lung lesion or lung cancer are excluded from this study.
* Patients not receiving care within the Baptist Memorial Healthcare Corporation are excluded from this study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Lung Cancer Patients coming through the Baptist health care system
Sampling Method: Non-Probability Sample
Enrollment: 781 (Actual)
Dates: Start 2014-10-09 (Actual); Primary Completion 2017-10-31 (Actual); Study Completion 2020-02-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Osarogiagbon, Principal Investigator — Baptist Memorial Health Care Corporation
Locations (1):
- Baptist Memorial Hospital, Memphis, Tennessee, United States

REFERENCES:
- [Derived] Shao H, Faris NR, Ward KD, Chen W, McHugh L, Smeltzer M, Ray MA, Osarogiagbon RU. Lung Cancer Patients' and Caregivers' Satisfaction With Multidisciplinary Versus Serial Care in a Community Healthcare Setting: A Prospective Comparative-Effectiveness Cohort Study. Clin Lung Cancer. 2023 Nov;24(7):e267-e274. doi: 10.1016/j.cllc.2023.06.006. Epub 2023 Jun 20. PMID 37451932
- [Derived] Smeltzer MP, Ray MA, Faris NR, Meadows-Taylor MB, Rugless F, Berryman C, Jackson B, Fehnel C, Pacheco A, McHugh L, Robbins ET, Ward KD, Klesges LM, Osarogiagbon RU. Prospective Comparative Effectiveness Trial of Multidisciplinary Lung Cancer Care Within a Community-Based Health Care System. JCO Oncol Pract. 2023 Jan;19(1):e15-e24. doi: 10.1200/OP.21.00815. Epub 2022 May 24. PMID 35609221
- [Derived] Smeltzer MP, Rugless FE, Jackson BM, Berryman CL, Faris NR, Ray MA, Meadows M, Patel AA, Roark KS, Kedia SK, DeBon MM, Crossley FJ, Oliver G, McHugh LM, Hastings W, Osborne O, Osborne J, Ill T, Ill M, Jones W, Lee HK, Signore RS, Fox RC, Li J, Robbins ET, Ward KD, Klesges LM, Osarogiagbon RU. Pragmatic trial of a multidisciplinary lung cancer care model in a community healthcare setting: study design, implementation evaluation, and baseline clinical results. Transl Lung Cancer Res. 2018 Feb;7(1):88-102. doi: 10.21037/tlcr.2018.01.02. PMID 29535915

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment process included a patient population of those receiving care and/or treatment for their lung cancer from physicians and clinics within the Baptist Cancer Center network, including sites in the Memphis metropolitan area, Oxford, Mississippi, and Jonesboro, Arkansas. Dates of recruitment were from October 2014 through May 2016.
Pre-assignment Details: Patient eligibility criteria: diagnosis of lung cancer within 6 weeks of screening date, an Eastern Cooperative Oncology Group (ECOG) performance status of 0-2, no previous lung cancer diagnosis, and no diagnosis of other cancers within the past 5 years. Caregivers and clinical care providers (doctors/nurses) of eligible patients also gave consent.
Groups:
- Multidisciplinary Clinic Patients: For the multidisciplinary arm, patients and their informal caregivers are seen by multiple specialists at a single appointment time.
- Serial Care Patients: For the serial care arm, matched serial care control patients receive the current system of linear, sequential, referral-based care delivery.
Period: Baseline Intervention
Arm/Group | Multidisciplinary Clinic Patients | Serial Care Patients | Multidisciplinary Caregivers | Serial Care Caregivers | Clinical Providers
Started | 178 | 348 | 100 | 144 | 11
Completed | 156 | 306 | 100 | 144 | 11
Not Completed | 22 | 42 | 0 | 0 | 0
Not completed — Death | 9 | 16 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 8 | 0 | 0 | 0
Not completed — Relocation | 2 | 0 | 0 | 0 | 0
Not completed — Out of window for initial survey | 6 | 13 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 5 | 0 | 0 | 0
Not completed — Other Disease | 3 | 0 | 0 | 0 | 0
Period: 3-month Follow up (Cumulative Counts)
Arm/Group | Multidisciplinary Clinic Patients | Serial Care Patients | Multidisciplinary Caregivers | Serial Care Caregivers | Clinical Providers
Started | 156 | 306 | 100 | 144 | 11 (Clinical providers received 6 month follow-up rather than 3 month follow-up at this stage.)
Completed | 99 | 189 | 50 | 62 | 8
Not Completed | 57 | 117 | 50 | 82 | 3
Not completed — Death | 33 | 57 | 0 | 0 | 0
Not completed — Lost to Follow-up | 2 | 7 | 50 | 82 | 3
Not completed — Withdrawal by Subject | 6 | 16 | 0 | 0 | 0
Not completed — Relocation | 0 | 1 | 0 | 0 | 0
Not completed — Out of window for follow-up survey | 16 | 36 | 0 | 0 | 0
Period: 6-month Follow up (Cumulative Counts)
Arm/Group | Multidisciplinary Clinic Patients | Serial Care Patients | Multidisciplinary Caregivers | Serial Care Caregivers | Clinical Providers
Started (Participants were able to complete a 6 month survey, even if they did not complete a 3 month survey.) | 156 | 306 | 100 | 144 | 8 (Clinical providers received 12 month follow-up rather than 6-month follow-up at this stage.)
Completed | 101 | 178 | 34 | 31 | 5
Not Completed | 55 | 128 | 66 | 113 | 3
Not completed — Death | 51 | 97 | 0 | 0 | 0
Not completed — Lost to Follow-up | 3 | 20 | 66 | 113 | 3
Not completed — Withdrawal by Subject | 1 | 9 | 0 | 0 | 0
Not completed — Relocation | 0 | 2 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Did not collect baseline information for caregivers or clinical providers since they were based on the patient information.
Groups:
- Multidisciplinary Clinic Patients: 150 multidisciplinary clinic patients and their informal caregivers are seen by multiple specialists at a single appointment time.
- Serial Care Patients: 300 matched serial care control patients who receive the current system of linear, sequential, referral-based care delivery.
- Total: Total of all reporting groups
Arm/Group | Multidisciplinary Clinic Patients | Serial Care Patients | Total
Number analyzed (Participants) | 178 | 348 | 526
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 55 | 147 | 202
  >=65 years | 123 | 201 | 324
Age, Continuous [Mean (Standard Deviation); unit: Years] | 68.85 (10.34) | 65.79 (9.62) | 66.83 (9.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 93 | 167 | 260
  Male | 85 | 181 | 266
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 3 | 12
  Not Hispanic or Latino | 164 | 308 | 472
  Unknown or Not Reported | 5 | 37 | 42
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 65 | 99 | 164
  White | 110 | 247 | 357
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 178 | 348 | 526
Primary Insurance [Count of Participants; unit: Participants]
  Medicare | 69 | 113 | 182
  Medicaid | 33 | 77 | 110
  Commercial | 66 | 147 | 213
  Self-insured/None | 10 | 11 | 21
Histology [Count of Participants; unit: Participants]
  Adenocarcinoma | 94 | 169 | 263
  Squamous Cell | 55 | 112 | 167
  Small Cell | 20 | 55 | 75
  Other | 9 | 12 | 21
ECOG [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group performance status scale. 0: fully active, able to carry on all pre-disease performance without restriction; 1: restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work; 2: ambulatory and capable of all self-care but unable to carry out any work activities, up and about more than 50% of waking hours; 3: capable of only limited self-care, confined to bed or chair more than 50% of waking hours; 4: completely disabled, cannot carry on any self-care; 5: dead.
  Participants
    0 | 80 | 118 | 198
    1 | 86 | 182 | 268
    2 | 12 | 43 | 55
    3 | 0 | 5 | 5
Initial Stage [Count of Participants; unit: Participants] — Initial Stage is the patient's clinical stage at initial lesion detection as determined by a radiologic scan that first showed a lesion. The staging reported uses the AJCC 7th edition Tumor/Node/Metastasis (TNM) framework for lung cancer staging. Lower staging (Stage IA) is considered a better prognosis than higher staging (Stage IV). For each stage, an earlier letter means a lower stage. Occult carcinoma means the main tumor can't be assessed. In this study, a change in clinical staging from initial to independently-calculated stage measures the impact of pre-treatment decision-making.
  Participants
    Stage I | 0 | 1 | 1
    Stage IA | 38 | 57 | 95
    Stage IB | 13 | 26 | 39
    Stage II | 0 | 1 | 1
    Stage IIA | 12 | 21 | 33
    Stage IIB | 11 | 22 | 33
    Stage IIIA | 48 | 62 | 110
    Stage IIIB | 17 | 24 | 41
    Stage IV | 39 | 132 | 171
    Occult Carcinoma | 0 | 2 | 2
Independently Calculated Clinical Stage [Count of Participants; unit: Participants] — Independently calculated clinical stage refers to the clinical stage immediately before the onset of first line treatment is determined. The independent calculation is performed by a trained research team member using all available pre-treatment clinical information and following the AJCC 7th edition Tumor/Node/Metastasis (TNM) guidelines for lung cancer. Lower staging (Stage 0) is considered a better prognosis than higher staging (Stage IV). Within each stage, an earlier letter means a lower stage.
  Participants
    Stage 0 | 0 | 1 | 1
    Stage IA | 36 | 57 | 93
    Stage IB | 13 | 24 | 37
    Stage IIA | 15 | 16 | 31
    Stage IIB | 13 | 14 | 27
    Stage IIIA | 33 | 56 | 89
    Stage IIIB | 16 | 28 | 44
    Stage IV | 52 | 152 | 204
Independently Calculated Clinical T Category [Count of Participants; unit: Participants] — The T category measures the size and extent of the primary tumor. Lower T categories (T1 tumor 3 cm or less) are considered better prognosis than higher T categories (T4 tumor larger than 7 cm, 2+ separate tumor nodules, or growth between the lungs). Independently calculated clinical T category refers to the method by which the T category immediately before onset of first line treatment is determined. The independent calculation is performed by a trained researcher using all available pre-treatment clinical information following the AJCC 7th edition framework for lung cancer staging.
  Participants
    T0 | 1 | 4 | 5
    T1a | 35 | 57 | 92
    T1b | 23 | 48 | 71
    T2a | 35 | 81 | 116
    T2b | 20 | 40 | 60
    T3 | 28 | 50 | 78
    T4 | 36 | 66 | 102
    Insufficient Records | 0 | 2 | 2
Independently Calculated Clinical N Category [Count of Participants; unit: Participants] — The N category measures the degree of cancer spread to nearby lymph nodes. Lower N categories (N0 the cancer has not spread to nearby lymph nodes) are considered better prognosis than higher N categories (N2 cancer spread to lymph nodes between the lungs). Independently calculated clinical N category refers to the method by which the N category immediately before onset of first line treatment is determined. The independent calculation is performed by a trained researcher using all available pre-treatment clinical information following the AJCC 7th edition framework for lung cancer staging.
  Participants
    N0 | 92 | 156 | 248
    N1 | 13 | 29 | 42
    N2 | 46 | 113 | 159
    N3 | 27 | 49 | 76
    Insufficient Records | 0 | 1 | 1
Independently Calculated Clinical M Category [Count of Participants; unit: Participants] — M category refers to the spread (metastasis) of the cancer to distant sites. Lower M categories (M0 no distant spread) are considered better prognosis than higher M categories (M1b spread outside the chest to distant organs such as liver, bones, or brain). Independently calculated clinical M category refers to the method by which the M category immediately before onset of first line treatment is determined. The independent calculation is performed by a trained researcher using all available pre-treatment clinical information following the AJCC 7th edition framework for lung cancer staging.
  Participants
    M0 | 126 | 196 | 322
    M1a | 14 | 33 | 47
    M1b | 38 | 119 | 157

OUTCOME MEASURES:

1. Primary Outcome: Thoroughness of Invasive Staging, Multidisciplinary (MD) vs Serial Care (SC)
Description: Number of patients with a test that provides tissue confirmation of the stage-defining lesion. Tests include a biopsy of any identified suspicious metastatic lesion or the primary lesion in the absence of any other suspicious lesion. 2 group comparison between Multidisciplinary Clinic Patients and Serial Care Patients.
Time Frame: From the time of a patient's positive lung cancer diagnosis, to the start of a patient's first-line of treatment, an average of 1-2 months
Population: All Specific Aim 3 patients (patients with histologically confirmed lung cancer (irrespective of histology) and an Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) from 0 (asymptomatic) to 2 (symptomatic but out of bed for >50% of the day)).
Measure: Count of Participants; unit: Participants
Groups:
- Multidisciplinary Clinic Patients: Patients seen and treated in the Multidisciplinary Clinic.
- Serial Care Patients: Patients seen and treated in the standard, sequential-referral-based environment of care.
Arm/Group | Multidisciplinary Clinic Patients | Serial Care Patients
Number analyzed (Participants) | 178 | 348
Participants
  Yes | 108 | 168
  No | 70 | 180
Statistical Analysis 1: Comparison: Multidisciplinary Clinic Patients vs Serial Care Patients; Test type: Superiority; p = 0.0007, Regression, Logistic — Conditional logistic regression adjusted for the matched study design, sex, age, and histology; Odds Ratio (OR) = 2.03, 95% CI 2-sided [1.35 to 3.06] — Odds ratio comparing Multidisciplinary Clinic patients with and without invasive stage confirmation (numerator=108/70) to Serial Care patients with and without invasive stage confirmation (denominator=168/180) after adjustment for matched study

2. Primary Outcome: Thoroughness of Invasive Mediastinal Staging, MD vs SC
Description: Number of patients with a test (i.e., biopsy) that provides tissue confirmation of the presence or absence of mediastinal nodal metastasis. 2 group comparison between Multidisciplinary Clinic Patients and Serial Care Patients.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Multidisciplinary Clinic Patients | Serial Care Patients
Number analyzed (Participants) | 178 | 348
Participants
  Yes | 91 | 126
  No | 87 | 222
Statistical Analysis 1: Comparison: Multidisciplinary Clinic Patients vs Serial Care Patients; Test type: Superiority; p = 0.0022, Regression, Logistic — Conditional logistic regression adjusted for the matched study design, sex, age, and histology; Odds Ratio (OR) = 1.87, 95% CI 2-sided [1.25 to 2.80] — Odds ratio comparing Multidisciplinary Clinic patients with and without invasive mediastinal staging (numerator=91/87) to Serial Care patients with and without mediastinal invasive staging (denominator=126/222) after adjustment for matched study

3. Primary Outcome: Thoroughness of Bi-Modal Staging Practice, MD vs SC
Description: Number of patients receiving two forms of staging tests (bi-modal staging). Bi-modal staging is defined as a CT scan plus any other type of radiologic scan or any biopsy. 2 group comparison between Multidisciplinary Clinic Patients and Serial Care Patients.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Multidisciplinary Clinic Patients | Serial Care Patients
Number analyzed (Participants) | 178 | 348
Participants
  Yes | 161 | 267
  No | 17 | 81
Statistical Analysis 1: Comparison: Multidisciplinary Clinic Patients vs Serial Care Patients; Test type: Superiority; p = 0.0004, Regression, Logistic — Conditional logistic regression adjusted for the matched study design, sex, age, and histology; Odds Ratio (OR) = 3.12, 95% CI 2-sided [1.67 to 5.85] — Odds ratio comparing Multidisciplinary Clinic patients with and without bi-modal staging (numerator=161/17) to Serial Care patients with and without bi-modal staging (denominator=267/81) after adjustment for matched study design

4. Primary Outcome: Thoroughness of Tri-Modal Staging Practice, MD vs SC
Description: Number of patients receiving three forms of staging tests (tri-modal staging). Tri-modal staging is defined as a CT scan plus any other type of radiologic scan plus any biopsy, or PET/CT plus any biopsy. 2 group comparison between Multidisciplinary Clinic Patients and Serial Care Patients.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Multidisciplinary Clinic Patients | Serial Care Patients
Number analyzed (Participants) | 178 | 348
Participants
  Yes | 99 | 132
  No | 79 | 216
Statistical Analysis 1: Comparison: Multidisciplinary Clinic Patients vs Serial Care Patients; Test type: Superiority; p < 0.0001, Regression, Logistic — Conditional logistic regression adjusted for the matched study design, sex, age, and histology; Odds Ratio (OR) = 2.25, 95% CI 2-sided [1.50 to 3.36] — Odds ratio comparing Multidisciplinary Clinic patients with and without tri-modal staging (numerator=99/79) to Serial Care patients with and without tri-modal staging (denominator=132/216) after adjustment for matched study design

5. Primary Outcome: Thoroughness of Invasive Staging, MD vs SC (Conference) vs SC (no Conference)
Description: Number of patients with a test that provides tissue confirmation of the stage-defining lesion. Tests include a biopsy of any identified suspicious metastatic lesion or the primary lesion in the absence of any other suspicious lesion.
  This measure compares 3 groups, instead of 2, because some patients in the serial care group were presented for discussion in a multidisciplinary thoracic oncology conference while still not being seen in the multidisciplinary clinic setting. Therefore, we split the serial care group in two in order to measure the potential impact of a multidisciplinary conference model, separate from the multidisciplinary clinic model.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Serial Care Patients Presented in Conference: Serial care patients who were presented in the multidisciplinary conference but not seen in the multidisciplinary clinic.
- Serial Care Patients Not Presented in Conference: Serial care patients who were not presented in the multidisciplinary conference.
Arm/Group | Multidisciplinary Clinic Patients | Serial Care Patients Presented in Conference | Serial Care Patients Not Presented in Conference
Number analyzed (Participants) | 178 | 76 | 272
Participants
  Yes | 108 | 46 | 122
  No | 70 | 30 | 150
Statistical Analysis 1: Comparison: Multidisciplinary Clinic Patients vs Serial Care Patients Not Presented in Conference; Test type: Superiority; p = 0.0366, Regression, Logistic — Conditional logistic regression adjusted for the matched study design, sex, age, and histology; Odds Ratio (OR) = 2.580, 95% CI 2-sided [1.665 to 3.996] — Odds ratio comparing Multidisciplinary Clinic patients with and without invasive staging (numerator=108/70) to Serial Care patients not in conference with and without invasive staging (denominator=122/150) after adjustment for matched study design
Statistical Analysis 2: Comparison: Serial Care Patients Presented in Conference vs Serial Care Patients Not Presented in Conference; Test type: Superiority; p = 0.0779, Regression, Logistic — Conditional logistic regression adjusted for the matched study design, sex, age, and histology; Odds Ratio (OR) = 2.621, 95% CI 2-sided [1.473 to 4.665] — Odds ratio comparing Serial Care patients in conference with and without invasive staging (numerator=46/30) to Serial Care patients not in conference with and without invasive staging (denominator=122/150) after adjustment for matched study design

6. Primary Outcome: Thoroughness of Invasive Mediastinal Staging, MD vs SC (no Conference) vs SC (Conference)
Description: Number of patients with a test (i.e., biopsy) that provides tissue confirmation of the presence or absence mediastinal nodal metastasis.
  This measure compares 3 groups, instead of 2, because some patients in the serial care group were presented for discussion in a multidisciplinary thoracic oncology conference while still not being seen in the multidisciplinary clinic setting. Therefore, we split the serial care group in two in order to measure the potential impact of a multidisciplinary conference model, separate from the multidisciplinary clinic model.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Multidisciplinary Clinic Patients | Serial Care Patients Presented in Conference | Serial Care Patients Not Presented in Conference
Number analyzed (Participants) | 178 | 76 | 272
Participants
  Yes | 91 | 40 | 86
  No | 87 | 36 | 186
Statistical Analysis 1: Comparison: Multidisciplinary Clinic Patients vs Serial Care Patients Not Presented in Conference; Test type: Superiority; p = 0.0703, Regression, Logistic — Conditional logistic regression adjusted for the matched study design, sex, age, and histology; Odds Ratio (OR) = 2.358, 95% CI 2-sided [1.536 to 3.621] — Odds ratio comparing Multidisciplinary Clinic patients with and without mediastinal staging (numerator=91/87) to Serial Care patients not in conference with and without mediastinal staging (denominator=86/186) after adjustment for matched study
Statistical Analysis 2: Comparison: Serial Care Patients Presented in Conference vs Serial Care Patients Not Presented in Conference; Test type: Superiority; p = 0.0631, Regression, Logistic — Conditional logistic regression adjusted for the matched study design, sex, age, and histology; Odds Ratio (OR) = 2.535, 95% CI 2-sided [1.446 to 4.444] — Odds ratio comparing Serial Care patients in conference with and without mediastinal staging (numerator=40/36) to Serial Care patients not in conference with and without mediastinal staging (denominator=86/186) after adjustment for matched study

7. Primary Outcome: Thoroughness of Bi-Modal Staging Practice, MD vs SC (Conference) vs SC (no Conference)
Description: Number of patients receiving two forms of staging tests (bi-modal staging). Bi-modal staging is defined as a CT scan plus any other type of radiologic scan or any biopsy.
  This measure compares 3 groups, instead of 2, because some patients in the serial care group were presented for discussion in a multidisciplinary thoracic oncology conference while still not being seen in the multidisciplinary clinic setting. Therefore, we split the serial care group in two in order to measure the potential impact of a multidisciplinary conference model, separate from the multidisciplinary clinic model.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Multidisciplinary Clinic Patients | Serial Care Patients Presented in Conference | Serial Care Patients Not Presented in Conference
Number analyzed (Participants) | 178 | 76 | 272
Participants
  Yes | 161 | 62 | 205
  No | 17 | 14 | 67
Statistical Analysis 1: Comparison: Multidisciplinary Clinic Patients vs Serial Care Patients Not Presented in Conference; Test type: Superiority; p = 0.0010, Regression, Logistic — Conditional logistic regression adjusted for the matched study design, sex, age, and histology; Odds Ratio (OR) = 3.191, 95% CI 2-sided [1.671 to 6.093] — Odds ratio comparing Multidisciplinary Clinic patients with and without bi-modal staging (numerator=161/17) to Serial Care patients not in conference with and without bi-modal staging (denominator=205/67) after adjustment for matched study
Statistical Analysis 2: Comparison: Serial Care Patients Presented in Conference vs Serial Care Patients Not Presented in Conference; Test type: Superiority; p = 0.1972, Regression, Logistic — Conditional logistic regression adjusted for the matched study design, sex, age, and histology; Odds Ratio (OR) = 1.103, 95% CI 2-sided [0.526 to 2.314] — Odds ratio comparing Serial Care patients in conference with and without bi-modal staging (numerator=62/14) to Serial Care patients not in conference with and without bi-modal staging (denominator=205/67) after adjustment for matched study

8. Primary Outcome: Thoroughness of Tri-Modal Staging Practice, MD vs SC (Conference) vs SC (no Conference)
Description: Number of patients receiving three forms of staging tests (tri-modal staging). Tri-modal staging is defined as a CT scan plus any other type of radiologic scan plus any biopsy, or PET/CT plus any biopsy.
  This measure compares 3 groups, instead of 2, because some patients in the serial care group were presented for discussion in a multidisciplinary thoracic oncology conference while still not being seen in the multidisciplinary clinic setting. Therefore, we split the serial care group in two in order to measure the potential impact of a multidisciplinary conference model, separate from the multidisciplinary clinic model.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Multidisciplinary Clinic Patients | Serial Care Patients Presented in Conference | Serial Care Patients Not Presented in Conference
Number analyzed (Participants) | 178 | 76 | 272
Participants
  Yes | 99 | 39 | 93
  No | 79 | 37 | 179
Statistical Analysis 1: Comparison: Multidisciplinary Clinic Patients vs Serial Care Patients Not Presented in Conference; Test type: Superiority; p = 0.0055, Regression, Logistic; Odds Ratio (OR) = 2.739, 95% CI 2-sided [1.785 to 4.203] — Odds ratio comparing Multidisciplinary Clinic patients with and without tri-modal staging (numerator=99/79) to Serial Care patients not in conference with and without tri-modal staging (denominator=93/179) after adjustment for matched study
Statistical Analysis 2: Comparison: Serial Care Patients Presented in Conference vs Serial Care Patients Not Presented in Conference; Test type: Superiority; p = 0.2572, Regression, Logistic — Conditional logistic regression adjusted for the matched study design, sex, age, and histology; Odds Ratio (OR) = 2.242, 95% CI 2-sided [1.287 to 3.905] — Odds ratio comparing Serial Care patients in conference with and without tri-modal staging (numerator=39/37) to Serial Care patients not in conference with and without tri-modal staging (denominator=93/179) after adjustment for matched study

9. Primary Outcome: Stage-Appropriateness Treatment Selection, MD vs SC
Description: Number of patients for whom appropriate treatment was given, as determined by the patients' clinical stage and treatment guidelines stipulated by the National Comprehensive Cancer Network (NCCN). 2 group comparison between Multidisciplinary Clinic Patients and Serial Care Patients.
  For Stage I or II: surgery (or radiation therapy with documented contraindication to surgery or patient refusal); for Stage III: chemotherapy and radiation therapy with or without surgery; for Stage IV: systemic therapy (or palliative care with documented patient refusal or contraindication to systemic therapy).
Time Frame: as for outcome 1
Population: Patients with a conference lung cancer who enrolled in the study who did not die, or leave the study before treatment, or did not refuse treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Multidisciplinary Clinic Patients | Serial Care Patients
Number analyzed (Participants) | 173 | 338
Participants
  Yes | 140 | 232
  No | 33 | 106
Statistical Analysis 1: Comparison: Multidisciplinary Clinic Patients vs Serial Care Patients; Test type: Superiority; p = 0.0045, Regression, Logistic — Conditional logistic regression adjusted for the matched study design, sex, age, and histology; Odds Ratio (OR) = 2.01, 95% CI 2-sided [1.24 to 3.25] — Odds ratio comparing MD patients with and without stage appropriate treatment (numerator=140/33) to SC patients with and without stage appropriate treatment (denominator=232/106) after adjustment for matched study

10. Primary Outcome: Stage-Appropriateness Treatment Selection, MD vs SC (Conference) vs SC (no Conference)
Description: Number of patients for whom appropriate treatment was given, as determined by the patients' clinical stage and treatment guidelines stipulated by the National Comprehensive Cancer Network (NCCN).
  For Stage I or II: surgery (or radiation therapy with documented contraindication to surgery or patient refusal); for Stage III: chemotherapy and radiation therapy with or without surgery; for Stage IV: systemic therapy (or palliative care with documented patient refusal or contraindication to systemic therapy).
  This measure compares 3 groups, instead of 2, because some patients in the serial care group were presented for discussion in a multidisciplinary thoracic oncology conference while still not being seen in the multidisciplinary clinic setting. Therefore, we split the serial care group in two in order to measure the potential impact of a multidisciplinary conference model, separate from the multidisciplinary clinic model.
Time Frame: as for outcome 1
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Multidisciplinary Clinic Patients | Serial Care Patients Presented in Conference | Serial Care Patients Not Presented in Conference
Number analyzed (Participants) | 173 | 73 | 265
Participants
  Yes | 140 | 58 | 174
  No | 33 | 15 | 91
Statistical Analysis 1: Comparison: Multidisciplinary Clinic Patients vs Serial Care Patients Not Presented in Conference; We examined treatment selection practices with or without MD care in a single healthcare system; Test type: Superiority; p = 0.0474, Regression, Logistic — Conditional logistic regression adjusted for the matched study design, sex, age, and histology; Odds Ratio (OR) = 2.249, 95% CI 2-sided [1.368 to 3.699] — Odds ratio comparing MD patients with and without stage appropriate treatment (numerator=140/33) to SC patients not in conference with and without stage appropriate treatment (denominator=174/91) after adjustment for matched study
Statistical Analysis 2: Comparison: Serial Care Patients Presented in Conference vs Serial Care Patients Not Presented in Conference; Test type: Superiority; p = 0.6353, Regression, Logistic — Conditional logistic regression adjusted for the matched study design, sex, age, and histology; Odds Ratio (OR) = 1.751, 95% CI 2-sided [0.910 to 3.370] — Odds ratio comparing SC patients in conference with and without stage appropriate treatment (numerator=58/15) to SC patients not in conference with and without stage appropriate treatment (denominator=174/91) after adjustment for matched study

11. Primary Outcome: Timeliness of Communication, MD vs SC(Conference)
Description: Number of patients for whom formal, verified communication of care management decisions was made to all team members (providers inside and outside the multidisciplinary program, patients and their care-givers) within 48 hours of a care recommendation being made. 2 group comparison between Multidisciplinary Clinic Patients and Serial Care Patients.
Time Frame: Within 48 hours of a documented care recommendation made through the multidisciplinary thoracic oncology program
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Groups:
- Overall Conference: All Patients presented in conference
Arm/Group | Multidisciplinary Clinic Patients | Serial Care Patients Presented in Conference | Overall Conference
Number analyzed (Participants) | 178 | 76 | 254
Participants
  Yes | 168 | 74 | 242
  No | 10 | 2 | 12

12. Primary Outcome: Concordance Rate for Initial Conference Recommendations, MD vs SC (Conference)
Description: Number of patients for whom all recommendations made at the initial multidisciplinary conference were completed. 2 group comparison between Multidisciplinary Clinic Patients and Serial Care Patients. Note that two patients (one from the MD arm and one from the SC arm) have died before receiving recommendations and therefore were not analyzed for this outcome.
Time Frame: From the time of a patient's positive lung cancer diagnosis, to the end of a patient's last line of treatment, an average of 1-2 months
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Groups:
- Serial Care Conference Patients: Serial care patients who were presented in the multidisciplinary conference but not seen in the multidisciplinary clinic.
Arm/Group | Multidisciplinary Clinic Patients | Serial Care Conference Patients
Number analyzed (Participants) | 177 | 75
Participants
  Yes | 140 | 45
  No | 37 | 30
Statistical Analysis 1: Comparison: Multidisciplinary Clinic Patients vs Serial Care Conference Patients; Test type: Superiority; p = 0.0014, Regression, Logistic — Conditional logistic regression adjusted for the matched study design, sex, age, and histology; Odds Ratio (OR) = 2.955, 95% CI 2-sided [1.520 to 5.747] — Odds ratio comparing MD patients with and without concordance to recommendations (numerator=140/37) to SC conference patients with and without concordance to recommendations (denominator=45/30) after adjustment for matched study design

13. Primary Outcome: Concordance Rate for Initial Conference Recommendation(s) With Prior Condition Met, MD vs SC (Conference)
Description: Number of patients for whom all initial conference recommendations were completed, excluding conditional recommendations for which the prior condition was not met. 2 group comparison between Multidisciplinary Clinic Patients and Serial Care Patients. Note that two patients (one from the MD arm and one from the SC arm) have died before receiving recommendations and therefore were not analyzed for this outcome.
  E.g., if a recommendation was to have a PET/CT and then a staging biopsy if the PET showed suspicious metastatic disease, the staging biopsy recommendation was excluded from the concordance measure if the PET/CT did not happen or was negative.
Time Frame: as for outcome 12
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Multidisciplinary Clinic Patients | Serial Care Conference Patients
Number analyzed (Participants) | 177 | 75
Participants
  Yes | 145 | 49
  No | 32 | 26
Statistical Analysis 1: Comparison: Multidisciplinary Clinic Patients vs Serial Care Conference Patients; Test type: Superiority; p = 0.0019, Regression, Logistic — Conditional logistic regression adjusted for the matched study design, sex, age, and histology; Odds Ratio (OR) = 3.093, 95% CI 2-sided [1.519 to 6.299] — Odds ratio comparing MD patients with and without concordance to recommendations (numerator=145/32) to SC conference patients with and without concordance to recommendations (denominator=49/26) after adjustment for matched study design

14. Primary Outcome: Concordance Rate for Any Conference Recommendation, MD vs SC (Conference)
Description: Number of patients for whom any initial conference recommendation was completed. 2 group comparison between Multidisciplinary Clinic Patients and Serial Care Patients. Note that two patients (one from the MD arm and one from the SC arm) have died before receiving recommendations and therefore were not analyzed for this outcome.
Time Frame: as for outcome 12
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Multidisciplinary Clinic Patients | Serial Care Conference Patients
Number analyzed (Participants) | 177 | 75
Participants
  Yes | 174 | 71
  No | 3 | 4
Statistical Analysis 1: Comparison: Multidisciplinary Clinic Patients vs Serial Care Conference Patients; Test type: Superiority; p = 0.0499, Regression, Logistic — Conditional logistic regression adjusted for the matched study design, sex, age, and histology; Odds Ratio (OR) = 40.892, 95% CI 2-sided [1.002 to 999.999] — Odds ratio comparing MD patients with and without concordance to recommendations (numerator=174/3) to SC conference patients with and without concordance to recommendations (denominator=71/4) after adjustment for matched study design

15. Primary Outcome: Overall Concordance Rate Using a Hierarchy of Initial Conference Recommendations, MD vs SC (Conference)
Description: Number of patients for whom the overall initial conference recommendation was completed. 2 group comparison between Multidisciplinary Clinic Patients and Serial Care Patients. Note that two patients (one from the MD arm and one from the SC arm) have died before receiving recommendations and therefore were not analyzed for this outcome.
  The hierarchy to rank recommendations, from highest priority to lowest, was (1) treatment, (2) staging, (3) diagnosis, (4) surveillance.
  If a patient had a treatment recommendation and it happened, he/she was concordant. If treatment was recommended and it did not happen, he/she was discordant. If no treatment recommendation was made, then concordance was measured by whether or not the staging recommendation was met. If no staging recommendation was made, then the diagnostic recommendation was given priority for a concordance measurement. If no diagnostic recommendation, then a surveillance recommendation was used to measure overall concordance.
Time Frame: as for outcome 12
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Multidisciplinary Clinic Patients | Serial Care Conference Patients
Number analyzed (Participants) | 177 | 75
Participants
  Yes | 158 | 60
  No | 19 | 15
Statistical Analysis 1: Comparison: Multidisciplinary Clinic Patients vs Serial Care Conference Patients; Test type: Superiority; p = 0.0263, Regression, Logistic — Conditional logistic regression adjusted for the matched study design, sex, age, and histology; Odds Ratio (OR) = 2.663, 95% CI 2-sided [1.123 to 6.319] — Odds ratio comparing MD patients with and without concordance to recommendations (numerator=158/19) to SC conference patients with and without concordance to recommendations (denominator=60/15) after adjustment for matched study design

16. Primary Outcome: Concordance Rate for Treatment Recommendations With Prior Recommendations Completed, MD vs SC (Conference)
Description: Number of patients for whom the treatment recommendation made at the initial conference presentation was completed, excluding any patient for whom prior recommendations (staging, diagnosis, surveillance) were not also completed. 2 group comparison between Multidisciplinary Clinic Patients and Serial Care Patients.
Time Frame: as for outcome 12
Population: Patients with a conference lung cancer who enrolled in the study who did not die, or leave the study before treatment, or did not refuse treatment excluding any patient for whom prior recommendations (staging, diagnosis, surveillance) were not also completed.
Measure: Count of Participants; unit: Participants
Arm/Group | Multidisciplinary Clinic Patients | Serial Care Conference Patients
Number analyzed (Participants) | 101 | 46
Participants
  Yes | 87 | 38
  No | 14 | 8
Statistical Analysis 1: Comparison: Multidisciplinary Clinic Patients vs Serial Care Conference Patients; Test type: Superiority; p = 0.1503, Regression, Logistic — Conditional logistic regression adjusted for the matched study design, sex, age, and histology; Odds Ratio (OR) = 2.566, 95% CI 2-sided [0.711 to 9.269] — Odds ratio comparing MD patients with and without concordance to recommendations (numerator=87/14) to SC conference patients with and without concordance to recommendations (denominator=38/8) after adjustment for matched study design

17. Primary Outcome: Baseline Patient Survey Response Rate, MD vs SC
Description: Number of patients who completed a baseline patient survey
Time Frame: Baseline
Population: Patients who were offered baseline surveys (all Specific Aim 3 patients)
Measure: Count of Participants; unit: Participants
Arm/Group | Multidisciplinary Clinic Patients | Serial Care Patients
Number analyzed (Participants) | 178 | 348
Participants
  Yes | 156 | 306
  No | 22 | 42

18. Primary Outcome: 3-month Patient Survey Response Rate, MD vs SC
Description: Number of patients who completed a 3-month survey
Time Frame: Within 30 days of 3 months after baseline survey administration
Population: Patients who were offered 3-month surveys.
Measure: Count of Participants; unit: Participants
Arm/Group | Multidisciplinary Clinic Patients | Serial Care Patients
Number analyzed (Participants) | 156 | 306
Participants
  Yes | 99 | 189
  No | 57 | 117

19. Primary Outcome: 6-Month Patient Survey Response Rate, MD vs SC
Description: Number of patients who completed a 6-month survey
Time Frame: Within 30 days of 6 months after baseline survey administration
Population: Patients who were offered 6-month surveys. Note that patients were offered a 6-month survey even if they did not complete a 3-month survey.
Measure: Count of Participants; unit: Participants
Arm/Group | Multidisciplinary Clinic Patients | Serial Care Patients
Number analyzed (Participants) | 156 | 306
Participants
  Yes | 101 | 178
  No | 55 | 128

20. Primary Outcome: Patient Survey Scores at Baseline, MD vs SC
Description: Scores from patient surveys that measure quality of life and satisfaction with care received at the time the baseline survey was taken.
  Overall quality of health care - satisfaction with overall quality of health care since lung cancer diagnosis; range: 0-4 (higher is better) Financial burden of care - assessment of financial burden of care; range: 3-6 (sum of 3 items, higher is worse) Treatment decision-making: Surgery/Radiation/Chemotherapy - each 1 item; satisfaction with treatment decision-making; range: 0-2 (0=patient controlled; 1=shared decision; 2-physician decision; closer to 1 is best) Satisfaction with treatment plan - satisfaction with overall treatment plan; range: 1-5 (sum of 2 items, higher is better) Treatment decision-making: family role - satisfaction with family role in treatment decision-making; range: 0-2 (0=patient controlled; 1=shared decision; 2-physician decision; closer to 1 is best) (descriptions continued in 3 month survey description)
Time Frame: Baseline
Population: Patients who completed baseline surveys.
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | Multidisciplinary Clinic Patients | Serial Care Patients
Number analyzed (Participants) | 156 | 306
scores on a scale
  Overall quality of health care | 3.28 (0.99) | 3.15 (0.98)
  Financial burden of care | 5.32 (1.07) | 5.23 (1.12)
  Treatment decision-making: Surgery | 0.92 (0.60) | 1.14 (0.66)
  Treatment decision-making: Radiation | 0.97 (0.64) | 1.10 (0.60)
  Treatment decision-making: Chemotherapy | 1.03 (0.66) | 1.01 (0.63)
  Satisfaction with treatment plan | 3.95 (1.54) | 4.31 (1.20)
  Treatment decision-making: Family role | 0.73 (0.56) | 0.69 (0.53)
  Satisfaction with quality of care | 16.05 (2.56) | 13.58 (3.19)
  Satisfaction with physician communication | 18.42 (2.86) | 18.49 (2.85)
  Satisfaction with nurse communication | 16.55 (2.75) | 16.71 (2.81)
  Overall team satisfaction | 11.69 (3.41) | 12.24 (3.39)
  Physical well-being | 24.90 (7.61) | 24.88 (6.99)
  Social well-being | 17.73 (5.23) | 18.32 (3.89)
  Functional well-being | 22.14 (7.33) | 22.05 (7.04)
  Emotional well-being | 24.23 (6.04) | 24.04 (6.00)
  Lung cancer specific QOL | 31.87 (5.52) | 32.25 (5.80)
  Total Summary Score FACTL | 121.00 (21.42) | 121.71 (21.10)
  Generic score FACTG | 89.16 (18.17) | 89.40 (17.73)
  Trial outcome index | 78.70 (16.19) | 79.17 (15.61)
  Depression | 4.44 (3.91) | 4.92 (4.08)
  Anxiety | 4.53 (4.08) | 5.03 (4.29)

21. Primary Outcome: Patient Survey Scores at 3 Months, MD vs SC
Description: Scores from patient surveys that measure quality of life and satisfaction with care received at the time the 3-month survey was taken.
  (continued from baseline) Satisfaction with quality of care - overall satisfaction with care received from all care team members; range: 0-18 (sum of 6 items, higher is better) Satisfaction with physician communication - overall satisfaction with physician communication; range: 0-21 (sum of 7 items, higher is better) Satisfaction with nurse communication - overall satisfaction with nurse communication; range: 0-18 (sum of 6 items, higher is better) Overall team satisfaction - CAHPS satisfaction with care from team as a whole; range: 0-15 (sum of 4 items, higher is better) Physical/Social/Functional well-being - health-related quality of life relating to physical/social/functional well-being; range 0-28 (each a sum of 7 items, higher is better) (description continues in 6 month survey description)
Time Frame: Within 30 days of 3 months after baseline survey administration
Population: Patients who completed 3-month surveys.
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | Multidisciplinary Clinic Patients | Serial Care Patients
Number analyzed (Participants) | 99 | 189
scores on a scale
  Overall quality of health care | 3.31 (0.89) | 3.30 (0.82)
  Financial burden of care | 5.25 (1.16) | 5.11 (1.19)
  Treatment decision-making: Surgery | 0.93 (0.61) | 1.17 (0.64)
  Treatment decision-making: Radiation | 1.07 (0.55) | 1.13 (0.66)
  Treatment decision-making: Chemotherapy | 0.97 (0.58) | 1.05 (0.53)
  Satisfaction with treatment plan | 4.60 (0.82) | 4.59 (0.84)
  Treatment decision-making: Family role | 0.72 (0.50) | 0.74 (0.47)
  Satisfaction with quality of care | 16.09 (2.36) | 14.33 (2.30)
  Satisfaction with physician communication | 19.03 (2.34) | 19.01 (2.10)
  Satisfaction with nurse communication | 17.17 (2.54) | 17.33 (1.73)
  Overall team satisfaction | 13.94 (2.04) | 13.69 (2.31)
  Physical well-being | 25.62 (7.00) | 26.25 (7.08)
  Social well-being | 18.42 (3.85) | 18.92 (3.25)
  Functional well-being | 22.57 (7.17) | 23.16 (6.55)
  Emotional well-being | 24.69 (5.50) | 24.85 (5.09)
  Lung cancer specific QOL | 33.31 (5.89) | 33.36 (5.06)
  Total Summary Score FACTL | 124.89 (22.12) | 126.59 (19.60)
  Generic score FACTG | 91.67 (18.33) | 93.16 (16.53)
  Trial outcome index | 81.39 (17.03) | 82.77 (15.14)
  Depression | 5.37 (4.15) | 4.81 (3.96)
  Anxiety | 4.79 (4.02) | 4.50 (4.01)

22. Primary Outcome: Patient Survey Scores at 6 Months, MD vs SC
Description: Scores from patient surveys that measure quality of life and satisfaction with care received at the time the 6-month survey was taken.
  (cont) Emotional well-being - health-related quality of life related to emotional well-being; range 0-30 (sum of 6 items, higher is better) Lung cancer specific QOL - health-related quality of life related to lung cancer diagnosis; range: 0-36 (sum of 9 items, higher is better) Total Summary Score FACTL - full survey, functional assessment of cancer therapy - lung; range: 0-136 (sum of 36 items, higher is better) Generic Score FACTG - full survey, functional assessment of cancer therapy - general; range: 0-108 (sum of 27 items, higher is better) Trial Outcome Index - health related quality of life - trial outcome index; range: 0-84 (sum of 23 items, higher is better) Depression/Anxiety - depression/anxiety measured by Hospital Anxiety and Depression Scale; range: 0-21 (sum of 7 items each, higher is worse)
Time Frame: Within 30 days of 6 months after baseline survey administration
Population: Patients who completed 6-month surveys.
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | Multidisciplinary Clinic Patients | Serial Care Patients
Number analyzed (Participants) | 101 | 178
scores on a scale
  Overall quality of health care | 3.36 (0.74) | 3.15 (0.87)
  Financial burden of care | 5.48 (0.99) | 5.06 (1.30)
  Treatment decision-making: Surgery | 1.15 (0.55) | 1.09 (0.58)
  Treatment decision-making: Radiation | 1.09 (0.62) | 1.05 (0.67)
  Satisfaction with treatment plan | 4.89 (0.46) | 4.58 (0.99)
  Treatment decision-making: Chemo | 1.15 (0.55) | 1.06 (0.61)
  Treatment decision-making: Family role | 0.83 (0.42) | 0.75 (0.54)
  Satisfaction with quality of care | 15.89 (2.21) | 14.41 (2.55)
  Satisfaction with physician communication | 19.33 (1.50) | 19.08 (1.85)
  Satisfaction with nurse communication | 17.32 (1.88) | 17.04 (2.27)
  Overall team satisfaction | 14.19 (1.59) | 13.73 (2.17)
  Physical well-being | 28.46 (5.59) | 26.94 (6.39)
  Social well-being | 18.62 (3.78) | 18.29 (3.80)
  Functional well-being | 24.22 (6.07) | 23.41 (6.54)
  Emotional well-being | 26.15 (4.63) | 25.26 (4.72)
  Lung cancer specific QOL | 34.49 (5.96) | 33.59 (5.74)
  Total Summary Score FACTL | 132.00 (18.26) | 128.00 (19.92)
  Generic score FACTG | 97.61 (14.19) | 94.26 (15.89)
  Trial outcome index | 86.92 (14.39) | 83.96 (15.56)
  Depression | 4.07 (3.31) | 4.81 (4.03)
  Anxiety | 3.99 (3.99) | 4.65 (3.72)

23. Primary Outcome: Baseline Caregiver Survey Response Rate, MD vs SC
Description: Number of caregivers who completed a baseline patient survey
Time Frame: Baseline
Population: Caregivers who completed surveys
Measure: Count of Participants; unit: Participants
Groups:
- Multidisciplinary Clinic Caregivers: Multidisciplinary clinic informal caregivers of patients who are seen by multiple specialists at a single appointment time.
- Serial Care Caregivers: Serial care control caregivers whose patients received the current system of linear, sequential, referral-based care delivery.
Arm/Group | Multidisciplinary Clinic Caregivers | Serial Care Caregivers
Number analyzed (Participants) | 100 | 144
Participants
  Yes | 100 | 144
  No | 0 | 0

24. Primary Outcome: 3-month Caregiver Survey Response Rate, MD vs SC
Description: Number of caregivers who completed a 3-month survey
Time Frame: Within 30 days of 3 months after baseline survey administration
Population: Caregivers who completed surveys
Measure: Count of Participants; unit: Participants
Arm/Group | Multidisciplinary Clinic Caregivers | Serial Care Caregivers
Number analyzed (Participants) | 100 | 144
Participants
  Yes | 50 | 62
  No | 50 | 82

25. Primary Outcome: 6-Month Caregiver Survey Response Rate, MD vs SC
Description: Number of caregivers who completed a 6-month survey
Time Frame: Within 30 days of 6 months after baseline survey administration
Population: Caregivers who completed surveys
Measure: Count of Participants; unit: Participants
Arm/Group | Multidisciplinary Clinic Caregivers | Serial Care Caregivers
Number analyzed (Participants) | 100 | 144
Participants
  Yes | 34 | 31
  No | 66 | 113

26. Primary Outcome: Caregiver Survey Scores at Baseline, MD vs SC
Description: Scores from caregiver surveys that measure quality of life and satisfaction with care received at the time the baseline survey was taken.
  Overall quality of health care - satisfaction with overall quality of health care since lung cancer diagnosis; range:0-4 (higher is better) Treatment decision-making: Surgery/Radiation/Chemotherapy - each 1 item; satisfaction with treatment decision-making; range: 0-2 (0=patient controlled; 1=shared decision; 2-physician decision; closer to 1 is best) Treatment decision-making: family role - satisfaction with family role in treatment decision-making; range: 0-2 (0=patient controlled; 1=shared decision; 2-physician decision; closer to 1 is best) Satisfaction with treatment plan - satisfaction with overall treatment plan; range: 0-2 (higher is better) Satisfaction patient can complete treatment plan; range: 0-2 (higher is better) (continued in 3 month survey description)
Time Frame: Baseline
Measure: Mean (Standard Error); unit: scores on a scale
Groups:
- Multidisciplinary Clinic Caregivers: Multidisciplinary clinic caregivers of patients seen by multiple specialists at a single appointment time.
- Serial Care Caregivers: Serial care control caregivers of patients who receive the current system of linear, sequential, referral-based care delivery.
Arm/Group | Multidisciplinary Clinic Caregivers | Serial Care Caregivers
Number analyzed (Participants) | 100 | 144
scores on a scale
  Overall quality of health care | 3.27 (0.98) | 3.14 (0.95)
  Treatment decision-making: Surgery | 0.78 (0.65) | 0.90 (0.71)
  Treatment decision-making: Radiation | 0.94 (0.69) | 1.03 (0.67)
  Treatment decision-making: Chemo | 0.88 (0.59) | 0.98 (0.63)
  Treatment decision-making: Family role | 0.68 (0.50) | 0.73 (0.52)
  Satisfaction with treatment plan | 1.40 (0.83) | 1.61 (0.66)
  Satisfaction patient can complete treatment plan | 1.44 (0.80) | 1.63 (0.68)
  Satisfaction with quality of care | 16.41 (2.57) | 13.90 (2.94)
  Satisfaction with physician communication | 18.95 (2.48) | 18.76 (2.52)
  Satisfaction with nurse communication | 21.96 (4.29) | 22.46 (3.68)
  Overall team satisfaction | 10.66 (2.29) | 10.57 (2.29)
  Depression | 3.12 (3.49) | 3.76 (3.45)
  Anxiety | 6.57 (4.45) | 6.90 (4.77)
  Physical Functioning QOL | 78.23 (27.38) | 77.24 (25.88)
  Physical health problems QOL | 74.49 (38.46) | 68.71 (42.04)
  Pain QOL | 81.89 (26.14) | 80.32 (28.98)
  General health perceptions | 72.13 (19.63) | 69.35 (21.04)
  Energy/Fatigue QOL | 57.66 (21.02) | 59.04 (20.62)
  Social Functioning QOL | 78.98 (26.60) | 76.97 (24.83)
  Emotional health problems QOL | 74.75 (40.15) | 72.77 (40.61)
  Emotional well-being QOL | 65.09 (22.96) | 68.33 (19.17)

27. Primary Outcome: Caregiver Survey Scores at 3 Months, MD vs SC
Description: Scores from caregiver surveys that measure quality of life and satisfaction with care received at the time the 3-month survey was taken.
  (cont) Satisfaction with quality of care - overall satisfaction with care received from all care team members; range: 0-18 (sum of 6 items, higher is better) Satisfaction with physician communication - overall satisfaction with physician communication; range: 0-28 (sum of 7 items, higher is better) Satisfaction with nurse communication - overall satisfaction with nurse communication; range: 6-24 (sum of 6 items, higher is better) Overall team satisfaction - CAHPS satisfaction with care from team as a whole; range: 0-15 (sum of 4 items, higher is better) Depression/Anxiety - depression/anxiety measured by Hospital Anxiety and Depression Scale; range: 0-21 (sum of 7 items, higher is worse) (continued in 6 month survey description)
Time Frame: Within 30 days of 3 months after baseline survey administration
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | Multidisciplinary Clinic Caregivers | Serial Care Caregivers
Number analyzed (Participants) | 50 | 62
scores on a scale
  Overall quality of health care | 3.32 (0.96) | 3.55 (0.67)
  Treatment decision-making: Surgery | 0.71 (0.69) | 1.08 (0.65)
  Treatment decision-making: Radiation | 0.90 (0.60) | 1.00 (0.58)
  Treatment decision-making: Chemo | 0.78 (0.64) | 1.13 (0.58)
  Treatment decision-making: Family role | 0.64 (0.53) | 0.75 (0.48)
  Satisfaction with treatment plan | 1.80 (0.49) | 1.81 (0.44)
  Satisfaction patient can complete treatment plan | 1.86 (0.42) | 1.89 (0.32)
  Satisfaction with quality of care | 16.82 (2.14) | 14.54 (2.38)
  Satisfaction with physician communication | 19.30 (1.63) | 19.22 (2.45)
  Satisfaction with nurse communication | 23.36 (1.66) | 23.28 (2.59)
  Overall team satisfaction | 11.52 (0.89) | 11.46 (1.13)
  Depression | 3.72 (3.10) | 3.04 (3.10)
  Anxiety | 6.20 (4.10) | 6.04 (5.05)
  Physical Functioning QOL | 76.92 (26.13) | 73.67 (27.78)
  Physical health problems QOL | 68.37 (38.79) | 63.43 (42.26)
  Pain QOL | 68.37 (38.79) | 63.43 (42.26)
  General health perceptions | 73.90 (20.16) | 69.14 (20.44)
  Energy/Fatigue QOL | 57.70 (18.30) | 58.30 (16.79)
  Social Functioning QOL | 73.60 (27.08) | 80.19 (23.03)
  Emotional health problems QOL | 62.67 (40.76) | 67.28 (43.19)
  Emotional well-being QOL | 68.37 (14.61) | 67.80 (20.82)

28. Primary Outcome: Caregiver Survey Scores at 6 Months, MD vs SC
Description: Scores from caregiver surveys that measure quality of life and satisfaction with care received at the time the 6-month survey was taken.
  (cont) Physical Functioning QOL - 10 items; Physical Health Problems QOL - 4 items; Pain QOL - 2 items; General health perceptions - 5 items; Energy/fatigue QOL - 4 items; Social Functioning QOL - 2 items; Emotional health problems QOL - 3 items; Emotional well-being QOL - 5 items.
  All health related quality of life measures are from the SF-36 survey tool, and use a range of 0-100 mean score (higher is better).
Time Frame: Within 30 days of 6 months after baseline survey administration
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | Multidisciplinary Clinic Caregivers | Serial Care Caregivers
Number analyzed (Participants) | 34 | 31
scores on a scale
  Overall quality of health care | 3.24 (0.87) | 3.23 (0.92)
  Treatment decision-making: Surgery | 1.05 (0.67) | 0.91 (0.70)
  Treatment decision-making: Radiation | 1.05 (0.83) | 0.88 (0.70)
  Treatment decision-making: Chemo | 1.03 (0.68) | 1.00 (0.71)
  Treatment decision-making: Family role | 0.78 (0.49) | 0.76 (0.54)
  Satisfaction with treatment plan | 1.79 (0.48) | 1.86 (0.35)
  Satisfaction patient can complete treatment plan | 1.78 (0.58) | 1.72 (0.57)
  Satisfaction with quality of care | 16.33 (2.20) | 14.14 (2.96)
  Satisfaction with physician communication | 19.27 (2.41) | 19.50 (1.44)
  Satisfaction with nurse communication | 22.88 (3.50) | 23.36 (1.71)
  Overall team satisfaction | 11.27 (1.42) | 11.73 (0.77)
  Depression | 2.97 (2.89) | 3.45 (2.91)
  Anxiety | 5.42 (3.67) | 5.23 (3.01)
  Physical Functioning QOL | 75.15 (28.84) | 79.67 (25.10)
  Physical health problems QOL | 73.48 (41.43) | 69.32 (46.25)
  Pain QOL | 81.44 (25.41) | 84.66 (28.85)
  General health perceptions | 74.09 (17.30) | 62.95 (21.31)
  Energy/Fatigue QOL | 59.75 (22.51) | 54.85 (15.39)
  Social Functioning QOL | 76.59 (24.15) | 80.91 (24.96)
  Emotional health problems QOL | 72.73 (40.36) | 74.24 (42.33)
  Emotional well-being QOL | 67.60 (18.43) | 63.33 (18.31)

29. Primary Outcome: Timeliness of Care, MD vs SC
Description: Aggregate time in days from enrollment to a specific care delivery endpoint including: from initial detection of lesion to initial biopsy, from initial detection to non-invasive staging, from initial detection to invasive staging, and from initial detection to definitive treatment. 2 group comparison between Multidisciplinary Clinic Patients and Serial Care Patients.
Time Frame: From the time of a patient's initial lesion detection to the designated step in the care process, as noted per row below
Population: Not every patient went to every step, therefore the times only include patients that completed that step.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Multidisciplinary Clinic Patients | Serial Care Patients
Number analyzed (Participants) | 178 | 348
Days
  From Initial detection of lesion to initial biopsy: number analyzed (Participants) | 123 | 207
  From Initial detection of lesion to initial biopsy | 25 [9 to 71] | 15 [4 to 40]
  From initial detection to non-invasive staging: number analyzed (Participants) | 169 | 301
  From initial detection to non-invasive staging | 20 [8 to 44] | 16 [3 to 40]
  From initial detection to invasive staging: number analyzed (Participants) | 93 | 136
  From initial detection to invasive staging | 29 [16 to 79] | 20 [6 to 61]
  From initial detection to definitive treatment: number analyzed (Participants) | 156 | 288
  From initial detection to definitive treatment | 60 [41 to 139] | 57 [33 to 93]
Statistical Analysis 1: Comparison: Multidisciplinary Clinic Patients vs Serial Care Patients; Time from Initial Detection of Lesion to Diagnostic Biopsy; Test type: Superiority; p = 0.0042, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Multidisciplinary Clinic Patients vs Serial Care Patients; Time from Initial Detection of Lesion to Non-invasive Staging Test; Test type: Superiority; p = 0.0805, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Multidisciplinary Clinic Patients vs Serial Care Patients; Time from Initial Detection of Lesion to Invasive Staging Test; Test type: Superiority; p = 0.0073, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Multidisciplinary Clinic Patients vs Serial Care Patients; Time from Initial Detection of Lesion to Definitive Treatment; Test type: Superiority; p = 0.0579, Wilcoxon (Mann-Whitney)

30. Primary Outcome: Timeliness of Care, MD vs SC (Conference) vs SC (no Conference)
Description: Aggregate time in days from enrollment to specific care delivery endpoint including: from initial detection of lesion to initial biopsy, from initial detection to non-invasive staging, from initial detection to invasive staging, and from initial detection to definitive treatment.
  This measure compares 3 groups, instead of 2, because some patients in the serial care group were presented for discussion in a multidisciplinary thoracic oncology conference while still not being seen in the multidisciplinary clinic setting. Therefore, we split the serial care group in two in order to measure the potential impact of a multidisciplinary conference model, separate from the multidisciplinary clinic model.
Time Frame: as for outcome 29
Population: Not every patient went to every step, therefore the times only include patients that completed that step.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Multidisciplinary Clinic Patients | Serial Care Patients Presented in Conference | Serial Care Patients Not Presented in Conference
Number analyzed (Participants) | 178 | 76 | 272
Days
  From Initial detection of lesion to initial biopsy: number analyzed (Participants) | 123 | 50 | 272
  From Initial detection of lesion to initial biopsy | 25 [9 to 71] | 18.5 [4 to 40] | 13 [4 to 40]
  From initial detection to non-invasive staging: number analyzed (Participants) | 169 | 67 | 272
  From initial detection to non-invasive staging | 20 [8 to 44] | 18 [6 to 40] | 16 [3 to 42]
  Initial detection of lesion to invasive staging: number analyzed (Participants) | 93 | 40 | 96
  Initial detection of lesion to invasive staging | 29 [16 to 79] | 40 [9 to 80] | 14 [5 to 48]
  From initial detection to definitive treatment: number analyzed (Participants) | 156 | 66 | 222
  From initial detection to definitive treatment | 60 [41 to 139] | 69 [44 to 160] | 54 [30 to 90]
Statistical Analysis 1: Comparison: Multidisciplinary Clinic Patients vs Serial Care Patients Presented in Conference vs Serial Care Patients Not Presented in Conference; Time from Initial Detection of Lesion to Diagnostic Biopsy; Test type: Superiority; p = 0.0146, Kruskal-Wallis
Statistical Analysis 2: Comparison: Multidisciplinary Clinic Patients vs Serial Care Patients Presented in Conference vs Serial Care Patients Not Presented in Conference; Time from Initial Detection of Lesion to Non-invasive Staging Test; Test type: Superiority; p = 0.16, Kruskal-Wallis
Statistical Analysis 3: Comparison: Multidisciplinary Clinic Patients vs Serial Care Patients Presented in Conference vs Serial Care Patients Not Presented in Conference; Time from Initial Detection of Lesion to Invasive Staging Test; Test type: Superiority; p = 0.0014, Kruskal-Wallis
Statistical Analysis 4: Comparison: Multidisciplinary Clinic Patients vs Serial Care Patients Presented in Conference vs Serial Care Patients Not Presented in Conference; Time from Initial Detection of Lesion to Definitive Treatment; Test type: Superiority; p = 0.0037, Kruskal-Wallis

31. Primary Outcome: Clinical Provider Survey Responses - Ease of Referring Patients to the Conference
Description: Responses from clinical providers will measure provider satisfaction and obstacles to institutional multidisciplinary care.
Time Frame: After a provider referred their 5th patient to the multidisciplinary conference (baseline), then within 30 days of 6 months and 12 months, respectively, after baseline survey was completed
Population: Any clinical provider who referred at least 5 patients to the multidisciplinary program and consented to take satisfaction surveys.
Measure: Count of Participants; unit: Participants
Groups:
- Baseline: Clinical providers who referred more than 5 patients to the multidisciplinary program
- 6 Month Follow up: 6-month follow up of clinical providers who referred more than 5 patients to the multidisciplinary program
- 12 Month Follow-up: 12 month follow up of clinical providers who referred more than 5 patients to the multidisciplinary program
Arm/Group | Baseline | 6 Month Follow up | 12 Month Follow-up
Number analyzed (Participants) | 11 | 8 | 5
Participants
  Very Satisfied | 9 | 7 | 5
  Satisfied | 2 | 1 | 0
  Somewhat satisfied | 0 | 0 | 0
  Somewhat dissatisfied | 0 | 0 | 0
  Dissatisfied | 0 | 0 | 0
  Very Dissatisfied | 0 | 0 | 0

32. Primary Outcome: Clinical Provider Survey Responses - How Quickly my Patients Get Scheduled to be Discussed at the Conference
Description: as for outcome 31
Time Frame: as for outcome 31
Population: as for outcome 31
Measure: Count of Participants; unit: Participants
Arm/Group | Baseline | 6 Month Follow up | 12 Month Follow-up
Number analyzed (Participants) | 11 | 8 | 5
Participants
  Very satisfied | 10 | 7 | 5
  Satisfied | 1 | 1 | 0
  Somewhat satisfied | 0 | 0 | 0
  Dissatisfied | 0 | 0 | 0
  Very Dissatisfied | 0 | 0 | 0

33. Primary Outcome: Clinical Provider Survey Responses - The Helpfulness of the Staff in Scheduling Patients
Description: as for outcome 31
Time Frame: as for outcome 31
Population: as for outcome 31
Measure: Count of Participants; unit: Participants
Arm/Group | Baseline | 6 Month Follow up | 12 Month Follow-up
Number analyzed (Participants) | 11 | 8 | 5
Participants
  Very Satisfied | 10 | 8 | 5
  Satisfied | 1 | 0 | 0
  Somewhat satisfied | 0 | 0 | 0
  Somewhat dissatisfied | 0 | 0 | 0
  Dissatisfied | 0 | 0 | 0
  Very Dissatisfied | 0 | 0 | 0

34. Primary Outcome: Clinical Provider Survey Responses - The Quality of Treatment Recommendations That I Received for my Patient
Description: as for outcome 31
Time Frame: as for outcome 31
Population: as for outcome 31
Measure: Count of Participants; unit: Participants
Arm/Group | Baseline | 6 Month Follow up | 12 Month Follow-up
Number analyzed (Participants) | 11 | 8 | 5
Participants
  Very Satisfied | 10 | 6 | 5
  Satisfied | 1 | 2 | 0
  Somewhat satisfied | 0 | 0 | 0
  Somewhat dissatisfied | 0 | 0 | 0
  Dissatisfied | 0 | 0 | 0
  Very Dissatisfied | 0 | 0 | 0

35. Primary Outcome: Clinical Provider Survey Responses - How Quickly I Receive Feedback on my Patient
Description: as for outcome 31
Time Frame: as for outcome 31
Population: as for outcome 31
Measure: Count of Participants; unit: Participants
Arm/Group | Baseline | 6 Month Follow up | 12 Month Follow-up
Number analyzed (Participants) | 11 | 8 | 5
Participants
  Very Satisfied | 10 | 7 | 5
  Satisfied | 1 | 1 | 0
  Somewhat satisfied | 0 | 0 | 0
  Dissatisfied | 0 | 0 | 0
  Very Dissatisfied | 0 | 0 | 0

36. Primary Outcome: Clinical Provider Survey Responses - The Consistency With Which my Patients Are Sent Back for Further Treatment
Description: as for outcome 31
Time Frame: as for outcome 31
Population: as for outcome 31
Measure: Count of Participants; unit: Participants
Arm/Group | Baseline | 6 Month Follow up | 12 Month Follow-up
Number analyzed (Participants) | 11 | 8 | 5
Participants
  Very Satisfied | 10 | 7 | 5
  Satisfied | 0 | 0 | 0
  Somewhat satisfied | 0 | 0 | 0
  Somewhat dissatisfied | 0 | 0 | 0
  Dissatisfied | 0 | 0 | 0
  Very Dissatisfied | 0 | 0 | 0
  N/A | 1 | 1 | 0

37. Primary Outcome: Patient Overall Survival
Description: Overall survival, defined as the time from cancer diagnosis to death from any cause or data censoring, is analyzed and summarized with the survival probabilities over time using the Kaplan-Meier method. Confidence intervals for the 1- and 3- year survival probabilities are reported. Additionally, the Cox proportional hazard model was used to estimate hazard ratios which are reported in the statistical analyses with 95% confidence intervals.
Time Frame: As measured from the time from cancer diagnosis to death or data censor, up to 6 years
Measure: Number (95% Confidence Interval); unit: survival probability
Arm/Group | Multidisciplinary Clinic Patients | Serial Care Patients
Number analyzed (Participants) | 178 | 348
survival probability
  1-year overall survival estimate | 0.58 [0.51 to 0.65] | 0.60 [0.54 to 0.65]
  3-year overall survival estimate | 0.34 [0.27 to 0.41] | 0.36 [0.31 to 0.41]
Statistical Analysis 1: Comparison: Multidisciplinary Clinic Patients vs Serial Care Patients; Test type: Superiority; p = 0.7506, Log Rank
Statistical Analysis 2: Comparison: Multidisciplinary Clinic Patients vs Serial Care Patients; Test type: Superiority; p = 0.54, Regression, Cox; Hazard Ratio (HR) = 1.08, 95% CI 2-sided [0.85 to 1.36] — Comparison is Multidisciplinary/Serial Care

38. Primary Outcome: Patient Overall Survival With SC Further Broken Down
Description: Overall survival, defined as the time from cancer diagnosis to death from any cause or data censoring, is analyzed and summarized with the survival probabilities over time using the Kaplan-Meier method. Confidence intervals for the 1- and 3- year survival probabilities are reported. Additionally, the Cox proportional hazard model was used to estimate hazard ratios which are reported in the statistical analyses with 95% confidence intervals.
  This measure compares 3 groups, instead of 2, because some patients in the serial care group were presented for discussion in a multidisciplinary thoracic oncology conference while still not being seen in the multidisciplinary clinic setting. Therefore, we split the serial care group in two in order to measure the potential impact of a multidisciplinary conference model, separate from the multidisciplinary clinic model.
Time Frame: As measured from the time from cancer diagnosis to death or data censor, up to 6 years
Measure: Number (95% Confidence Interval); unit: survival probability
Arm/Group | Multidisciplinary Clinic Patients | Serial Care Patients Presented in Conference | Serial Care Patients Not Presented in Conference
Number analyzed (Participants) | 178 | 76 | 272
survival probability
  1-year overall survival estimate | 0.58 [0.51 to 0.65] | 0.64 [0.53 to 0.74] | 0.58 [0.52 to 0.64]
  3-year overall survival estimate | 0.34 [0.27 to 0.41] | 0.41 [0.30 to 0.52] | 0.34 [0.29 to 0.40]
Statistical Analysis 1: Comparison: Multidisciplinary Clinic Patients vs Serial Care Patients Presented in Conference vs Serial Care Patients Not Presented in Conference; Test type: Superiority; p = 0.4847, Log Rank
Statistical Analysis 2: Comparison: Multidisciplinary Clinic Patients vs Serial Care Patients Not Presented in Conference; Test type: Superiority; p = 0.51, Regression, Cox; Hazard Ratio (HR) = 1.12, 95% CI 2-sided [0.87 to 1.43] — Comparison is Multidisciplinary/Serial Care Patients Not Presented in Conference
Statistical Analysis 3: Comparison: Serial Care Patients Presented in Conference vs Serial Care Patients Not Presented in Conference; Test type: Superiority; p = 0.51, Regression, Cox; Hazard Ratio (HR) = 1.19, 95% CI 2-sided [0.84 to 1.67] — Comparison is Serial Care Patients Presented in Conference/Serial Care Patients Not Presented in Conference

39. Primary Outcome: Patient Disease/Progression Free Survival
Description: Event-free survival (EFS), as measured from the time from cancer diagnosis to disease progression, death, or data censoring, is analyzed and summarized with the survival probabilities over time using the Kaplan-Meier method. Confidence intervals for the 1- and 3- year survival probabilities are reported. Additionally, the Cox proportional hazard model was used to estimate hazard ratios which are reported in the statistical analyses with 95% confidence intervals.
Time Frame: measured from the time from cancer diagnosis to disease progression, death, or data censoring, up to 6 years
Measure: Number (95% Confidence Interval); unit: survival probability
Arm/Group | Multidisciplinary Clinic Patients | Serial Care Patients
Number analyzed (Participants) | 178 | 348
survival probability
  1-year EFS survival estimate | 0.45 [0.38 to 0.53] | 0.48 [0.43 to 0.53]
  3-year EFS survival estimate | 0.26 [0.20 to 0.33] | 0.26 [0.21 to 0.31]
Statistical Analysis 1: Comparison: Multidisciplinary Clinic Patients vs Serial Care Patients; Test type: Superiority; p = 0.9874, Log Rank
Statistical Analysis 2: Comparison: Multidisciplinary Clinic Patients vs Serial Care Patients; Test type: Superiority; p = 0.80, Regression, Cox; Hazard Ratio (HR) = 1.03, 95% CI 2-sided [0.82 to 1.29] — Comparison is Multidisciplinary/Serial Care

40. Primary Outcome: Patient Disease/Progression Free Survival With SC Further Broken Down
Description: Event-free survival (EFS), as measured from the time from cancer diagnosis to disease progression, death, or data censoring, is analyzed and summarized with the survival probabilities over time using the Kaplan-Meier method. Confidence intervals for the 1- and 3- year survival probabilities are reported. Additionally, the Cox proportional hazard model was used to estimate hazard ratios which are reported in the statistical analyses with 95% confidence intervals.
  This measure compares 3 groups, instead of 2, because some patients in the serial care group were presented for discussion in a multidisciplinary thoracic oncology conference while still not being seen in the multidisciplinary clinic setting. Therefore, we split the serial care group in two in order to measure the potential impact of a multidisciplinary conference model, separate from the multidisciplinary clinic model.
Time Frame: As measured from the time from cancer diagnosis to death or data censor, up to 6 years
Measure: Number (95% Confidence Interval); unit: survival probability
Arm/Group | Multidisciplinary Clinic Patients | Serial Care Patients Presented in Conference | Serial Care Patients Not Presented in Conference
Number analyzed (Participants) | 178 | 76 | 272
survival probability
  1-year EFS survival estimate | 0.45 [0.38 to 0.53] | 0.55 [0.43 to 0.65] | 0.46 [0.40 to 0.52]
  3-year EFS survival estimate | 0.26 [0.20 to 0.33] | 0.32 [0.22 to 0.43] | 0.24 [0.19 to 0.29]
Statistical Analysis 1: Comparison: Multidisciplinary Clinic Patients vs Serial Care Patients Presented in Conference vs Serial Care Patients Not Presented in Conference; Test type: Superiority; p = 0.5377, Log Rank
Statistical Analysis 2: Comparison: Multidisciplinary Clinic Patients vs Serial Care Patients Not Presented in Conference; Test type: Superiority; p = 0.73, Regression, Cox; Hazard Ratio (HR) = 1.06, 95% CI 2-sided [0.83 to 1.34] — Comparison is Multidisciplinary/Serial Care Patients Not Presented in Conference
Statistical Analysis 3: Comparison: Serial Care Patients Presented in Conference vs Serial Care Patients Not Presented in Conference; Test type: Superiority; p = 0.73, Regression, Cox; Hazard Ratio (HR) = 1.13, 95% CI 2-sided [0.82 to 1.57] — Comparison is Serial Care Patients Presented in Conference/Serial Care Patients Not Presented in Conference

ADVERSE EVENTS:
Time Frame: All-cause mortality for patients included a median follow up time of at least 1.5 years, up to 6 years in total.
Description: All-cause mortality was defined as the occurrence of death due to any cause. All-cause mortality for caregivers and clinical providers were not monitored.
  Serious and Other (Not Including Serious) Adverse Events were not monitored or assessed for patients, caregivers, or clinical providers.
  All-cause mortality reported is beyond the initial 6 month period noted in the participant flow table.
Arm/Group | Multidisciplinary Clinic Patients | Serial Care Patients
All-Cause Mortality (participants affected / at risk) | 125/178 | 239/348
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (5):
  • Statistical Analysis Plan (2015-03-09): https://cdn.clinicaltrials.gov/large-docs/97/NCT02123797/SAP_000.pdf
  • Informed Consent Form: Patient ICF (2016-11-10): https://cdn.clinicaltrials.gov/large-docs/97/NCT02123797/ICF_001.pdf
  • Informed Consent Form: Care Giver ICF (2016-11-10): https://cdn.clinicaltrials.gov/large-docs/97/NCT02123797/ICF_002.pdf
  • Informed Consent Form: Provider ICF (2016-11-10): https://cdn.clinicaltrials.gov/large-docs/97/NCT02123797/ICF_003.pdf
  • Study Protocol (2015-03-09): https://cdn.clinicaltrials.gov/large-docs/97/NCT02123797/Prot_004.pdf